CLINICAL TRIAL: NCT01711840
Title: Symbicort Turbuhaler 30/60 Clinical Experience Investigation for Treatment With Symbicort as Maintenance Therapy and as Needed in Response to Symptoms
Brief Title: Clinical Experience Investigation of Symbicort Turbuhaler as Maintenance Therapy and Reliever Therapy
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D589LL00001
Record Dates: First submitted 2012-10-19; First posted 2012-10-22 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Bronchial Asthma
Keywords: Bronchial asthma; Symbicort Turbuhaler
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Symbicort

SUMMARY:
The purpose of the investigation is to confirm the safety of patients receiving Symbicort Turbuhaler as maintenance and reliever therapy ( Symbicort SMART) under the post-marketing actual use.

DETAILED DESCRIPTION:
Symbicort Turbuhaler 30/60 Clinical Experience Investigation for treatment with Symbicort as maintenance therapy and as needed in response to symptoms

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving Symbicort Turbuhaler as maintenance and reliever therapy for the first time due to 'bronchial asthma ',and possibly requiring as-needed inhalations during the observation period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving Symbicort Turbuhaler as maintenance and reliever therapy for the first time due to 'bronchial asthma ',and possibly requiring as-needed inhalations during the observation period
Sampling Method: Non-Probability Sample
Enrollment: 2409 (Actual)
Dates: Start 2012-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Adverse event incidence | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Yoshida, MD, Study Director — AstraZeneca KK
Locations (47):
- Japan (47):
  - Research Site, Aichi, D589ll00001
  - Research Site, Akita, D589ll00001
  - Research Site, Aomori, D589ll00001
  - Research Site, Chiba, D589ll00001
  - Research Site, Ehime, D589ll00001
  - Research Site, Fukui, D589ll00001
  - Research Site, Fukuoka, D589ll00001
  - Research Site, Fukushima, D589ll00001
  - Research Site, Gifu, D589ll00001
  - Research Site, Gunma, D589ll00001
  - Research Site, Hiroshima, D589ll00001
  - Research Site, Hokkaido, D589ll00001
  - Research Site, Hyōgo, D589ll00001
  - Research Site, Ibaraki, D589ll00001
  - Research Site, Ishikawa, D589ll00001
  - Research Site, Kagawa, D589ll00001
  - Research Site, Kagoshima, D589ll00001
  - Research Site, Kanagawa, D589ll00001
  - Research Site, Kochi, D589ll00001
  - Research Site, Kumamoto, D589ll00001
  - Research Site, Kyoto, D589ll00001
  - Research Site, Mie, D589ll00001
  - Research Site, Miyagi, D589ll00001
  - Research Site, Miyazaki, D589ll00001
  - Research Site, Nagano, D589ll00001
  - Research Site, Nagasaki, D589ll00001
  - Research Site, Nara, D589ll00001
  - Research Site, Niigata, D589ll00001
  - Research Site, Numakunai, D589ll00001
  - Research Site, Okayama, D589ll00001
  - Research Site, Okinawa, D589ll00001
  - Research Site, Osaka, D589ll00001
  - Research Site, Ōita, D589ll00001
  - Research Site, Saga, D589ll00001
  - Research Site, Saitama, D589ll00001
  - Research Site, Shiga, D589ll00001
  - Research Site, Shimane, D589ll00001
  - Research Site, Shizuoka, D589ll00001
  - Research Site, Tochigi, D589ll00001
  - Research Site, Tokushima, D589ll00001
  - Research Site, Tokyo, D589ll00001
  - Research Site, Tottori, D589ll00001
  - Research Site, Toyama, D589ll00001
  - Research Site, Wakayama, D589ll00001
  - Research Site, Yamagata, D589ll00001
  - Research Site, Yamaguchi, D589ll00001
  - Research Site, Yamanashi, D589ll00001

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=550&filename=SynopsisD589LL00001.pdf